CLINICAL TRIAL: NCT01520727
Title: A Single Oral Ascending Dose Study to Investigate the Safety, Pharmacokinetics and Catechol-O-methyltransferase (COMT) Inhibition Profiles of BIA 9-1067 in Healthy Male Subjects
Brief Title: A Single Oral Ascending Dose Study of BIA 9-1067 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-101
Record Dates: First submitted 2012-01-18; First posted 2012-01-30 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson Disease
Keywords: BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; entacapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- BIA 9-1067 10 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 10 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 25 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 25 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 50 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 50 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 100 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 100 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 200 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 200 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 400 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 400 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 800 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 800 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 1200 mg (Experimental): BIA 9-1067 (Opicapone, OPC) - 1200 mg
  Interventions: Drug: BIA 9-1067
- Placebo (Placebo Comparator): Placebo (PLC): single-dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 9-1067 — single ascending doses in up to 8 sequential groups of 8 healthy young male subjects
  Other Names: Entacapone
  Arms: BIA 9-1067 10 mg; BIA 9-1067 100 mg; BIA 9-1067 1200 mg; BIA 9-1067 200 mg; BIA 9-1067 25 mg; BIA 9-1067 400 mg; BIA 9-1067 50 mg; BIA 9-1067 800 mg
Drug: Placebo — single-dose
  Arms: Placebo

SUMMARY:
The purpose of this study was to investigate the safety, tolerability, pharmacokinetics and catechol-O-methyltransferase (COMT) activity of BIA 9-1067 in healthy male subjects after single oral ascending doses.

DETAILED DESCRIPTION:
Single centre, randomised, double-blind, placebo-controlled study of single ascending doses in up to 8 sequential groups of 8 healthy young male subjects.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form before any study-specific screening procedure was performed.
* Aged between 18 and 45 years, inclusive.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead ECG.
* Non-smoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Exclusion Criteria:

* Any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, dermatological, haematological, neurologic, or psychiatric disease.
* Acute disease state (e.g., nausea, vomiting, fever, diarrhoea) within 7 days before study day 1.
* History of drug abuse within 1 year before study day 1.
* History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g
* Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
* Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA [3,4-methylenedioxy-methamphetamine; ecstasy]).
* History of any clinically important drug allergy.
* Prohibited Treatments: use of any investigational drug within 90 days or prescription drug within 30 days before investigational medical product (IMP) administration.
* Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 24 hours before study day 1.
* Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before IMP administration.
* Donation of blood (i.e. 450 mL) within 60 days before study day 1

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Fauchoux, MD, Principal Investigator — Biotrial
Locations (1):
- BIOTRIAL, Rennes, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIA 9-1067 10 mg | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | BIA 9-1067 200 mg | BIA 9-1067 400 mg | BIA 9-1067 800 mg | BIA 9-1067 1200 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067 10 mg | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | BIA 9-1067 200 mg | BIA 9-1067 400 mg | BIA 9-1067 800 mg | BIA 9-1067 1200 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 64
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 64

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs)
Description: Safety was evaluated from the number of reported adverse events (AEs)
Time Frame: 7 weeks
Measure: Number; unit: Number of Adverse Events
Arm/Group | BIA 9-1067 10 mg | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | BIA 9-1067 200 mg | BIA 9-1067 400 mg | BIA 9-1067 800 mg | BIA 9-1067 1200 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16
Number of Adverse Events | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 4

2. Secondary Outcome: Cmax - BIA 9-1067
Description: Cmax - maximum plasma concentration
Time Frame: pre-dose then post-dose. Hour 0.25, 0.5, 0,75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48 , 60 and 72 hours post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BIA 9-1067 10 mg | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | BIA 9-1067 200 mg | BIA 9-1067 400 mg | BIA 9-1067 800 mg | BIA 9-1067 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 130.7 (68.0) | 308.5 (128.1) | 522.2 (186.7) | 927.2 (378.9) | 1287.5 (585.6) | 2013.3 (608.7) | 2786.7 (1335.9) | 4883.3 (1501.5)

3. Secondary Outcome: Time to Cmax (Tmax)
Time Frame: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | BIA 9-1067 10 mg | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | BIA 9-1067 200 mg | BIA 9-1067 400 mg | BIA 9-1067 800 mg | BIA 9-1067 1200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 2.5 [2.0 to 4.0] | 1.5 [1.0 to 4.0] | 3.5 [1.5 to 4.0] | 1.8 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.5 to 5.0] | 2.5 [0.8 to 5.3] | 1.5 [1.0 to 3.0]

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 10 mg | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | BIA 9-1067 200 mg | BIA 9-1067 400 mg | BIA 9-1067 800 mg | BIA 9-1067 1200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 1/16
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/6 | 0/6 | 1/6 | 1/6 | 0/6 | 1/6 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIA 9-1067 10 mg (N=6) | BIA 9-1067 25 mg (N=6) | BIA 9-1067 50 mg (N=6) | BIA 9-1067 100 mg (N=6) | BIA 9-1067 200 mg (N=6) | BIA 9-1067 400 mg (N=6) | BIA 9-1067 800 mg (N=6) | BIA 9-1067 1200 mg (N=6) | Placebo (N=16)
Spastic Paraplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 10 mg (N=6) | BIA 9-1067 25 mg (N=6) | BIA 9-1067 50 mg (N=6) | BIA 9-1067 100 mg (N=6) | BIA 9-1067 200 mg (N=6) | BIA 9-1067 400 mg (N=6) | BIA 9-1067 800 mg (N=6) | BIA 9-1067 1200 mg (N=6) | Placebo (N=16)
Syncope Vasovagal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other